CLINICAL TRIAL: NCT06646913
Title: Transcutaneous Electrical Nerve Stimulation in Scleroderma
Brief Title: TENS in Scleroderma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Dinesh Khanna, MD, MS, Professor of Rheumatology, University of Michigan Scleroderma Program Director, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HUM00246152
Record Dates: First submitted 2024-10-04; First posted 2024-10-17 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Scleroderma; Gastroparesis; Systemic Sclerosis (SSc)
Keywords: TENS; Scleroderma; Gastroparesis; Pilot Study; Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse; Gastroparesis; Scleroderma, Systemic | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Scleroderma Patients with Gastroparesis Symptoms (Experimental)
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation — Patients will utilize the TENS device for 45 minutes, two times per day for the 4 week treatment period.
  Other Names: TENS

SUMMARY:
The goal of this pilot study is to assess the acceptability of the transcutaneous electrical acustimulation (TEA) device in treating Scleroderma-related gastroparesis. The main objective is:

To evaluate the acceptability of TEA as an intervention for alleviating symptoms of distension and bloating in individuals diagnosed with Scleroderma.

Participants will be provided with the TEA devices that will be applied to the skin for a total of 45 minutes twice daily after meals. Participants will be asked to fill out both daily diaries and biweekly questionnaires to assess for improvement in the gastroparesis symptoms. Participants will also be asked to complete the daily diaries in addition weekly questionnaires during a 4 week post-treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Classification of Systemic Sclerosis according to the 2013 American College of Rheumatology and European League against Rheumatism classification criteria.
2. Age >= 18 years
3. English speaking.
4. Participants who report moderate to severe symptoms of distension/bloating on UCLA Scleroderma Clinical Trials Consortium Gastrointestinal Tract Instrument 2.0
5. Stable GI specific therapy including prokinetics over the last 4 weeks.

Exclusion Criteria:

1. Pregnancy, or currently lactating.
2. A history of major abdominal surgery (other than cholecystectomy, appendectomy, or deemed as non-major by the investigators)
3. Unrelated active disorder which may involve abdominal pain, such as inflammatory bowel disease, diabetes or unstable thyroid disease.
4. Known allergy to adhesive ECG electrodes.
5. Known contraindications to TEA (e.g., cardiac pacemaker, epilepsy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Tolerability of the TENS device | 14 months
  1. Proportion of subjects who are able to complete the trial
  2. Proportion of subjects who utilize the device for at least 80% of the proposed applications.

SECONDARY OUTCOMES:
Efficacy of TENS in treating Scleroderma-related Gastroparesis | 14 months
  To assess the mean change in the GCSI Total score (0-4 where higher score reflects greater severity) after the TENS intervention.
Assessment of the Effect of TENS of Gastroparesis Symptoms | 14 months
  To assess the mean change in the GIT 2.0 Distention/Bloating scale (0-3.0 where 0 is lower severity and 3.0 is greater severity) after the TENS intervention.
Assessment of the Safety of TENS in Treating Scleroderma-related Gastroparesis | 14 months
  To evaluate the number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Revicki DA, Camilleri M, Kuo B, Norton NJ, Murray L, Palsgrove A, Parkman HP. Development and content validity of a gastroparesis cardinal symptom index daily diary. Aliment Pharmacol Ther. 2009 Sep 15;30(6):670-80. doi: 10.1111/j.1365-2036.2009.04078.x. Epub 2009 Jun 25. PMID 19558608
- [Background] Khanna D, Hays RD, Maranian P, Seibold JR, Impens A, Mayes MD, Clements PJ, Getzug T, Fathi N, Bechtel A, Furst DE. Reliability and validity of the University of California, Los Angeles Scleroderma Clinical Trial Consortium Gastrointestinal Tract Instrument. Arthritis Rheum. 2009 Sep 15;61(9):1257-63. doi: 10.1002/art.24730. PMID 19714600
- [Background] McMahan ZH, Kulkarni S, Chen J, Chen JZ, Xavier RJ, Pasricha PJ, Khanna D. Systemic sclerosis gastrointestinal dysmotility: risk factors, pathophysiology, diagnosis and management. Nat Rev Rheumatol. 2023 Mar;19(3):166-181. doi: 10.1038/s41584-022-00900-6. Epub 2023 Feb 6. PMID 36747090
- [Background] Song G, Trujillo S, Fu Y, Shibi F, Chen J, Fass R. Transcutaneous electrical stimulation for gastrointestinal motility disorders. Neurogastroenterol Motil. 2023 Nov;35(11):e14618. doi: 10.1111/nmo.14618. Epub 2023 Jun 8. PMID 37288650